CLINICAL TRIAL: NCT00371774
Title: Amevive Wisdom Acquired From Real-Time Evidence (A.W.A.R.E™) Program
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CA-08; NCT00214799 (obsolete NCT alias)
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; Plaque Psoriasis; Amevive®; alefacept
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Dermatologic patients in Canada for which Amevive is clinically indicated

SUMMARY:
Purpose:

To develop a real time national clinical database to support and share best practices,

1. To generate hypotheses for future clinical research
2. To understand how AMEVIVE is used in routine clinical practice/real world setting.

Each patient visit will include the following observational endpoints:

1. AMEVIVE dosing
2. Number of courses
3. Concomitant treatment
4. Response to treatment (patient and physician global assessments)
5. Status of other psoriasis-related medical conditions
6. Time to re-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Amevive is clinically indicated for the patient

Exclusion Criteria:

* Amevive is contraindicated for the patient

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Dermatologic patients in Canada
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2005-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Understand how AMEVIVE is used in routine clinical practice/real world setting | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Canada, Inc.
Locations (22):
- Canada (22):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - Saint John, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Barrie, Ontario
  - Concord, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - Markham, Ontario
  - Oakville, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Sainte-Foy, Quebec

REFERENCES:
- [Background] Searles G, Bissonnette R, Landells I, Shear NH. Preface: real-world clinical experience with alefacept-the Amevive Wisdom Acquired from Real-World Evidence (AWARE) study. J Cutan Med Surg. 2009 Dec;13 Suppl 3:S107-12. doi: 10.2310/7750.2009.00028. No abstract available. PMID 20053322
- [Background] Bissonnette R, Searles G, Landells I, Shear NH, Papp K, Lui H, Gulliver WP, Lynde C. The AWARE study: methodology and baseline characteristics. J Cutan Med Surg. 2009 Dec;13 Suppl 3:S113-21. doi: 10.2310/7750.2009.00029. PMID 20053323
- [Background] Landells I, Searles G, Bissonnette R, Shear NH, Vender R, Lui H. Efficacy outcomes in patients using alefacept in the AWARE study. J Cutan Med Surg. 2009 Dec;13 Suppl 3:S122-30. doi: 10.2310/7750.2009.00030. PMID 20053324
- [Background] Searles G, Bissonnette R, Landells I, Shear NH, Papp K, Lui H. Patterns of combination therapy with alefacept for the treatment of psoriasis in Canada in the AWARE study. J Cutan Med Surg. 2009 Dec;13 Suppl 3:S131-8. doi: 10.2310/7750.2009.00031. PMID 20053325
- [Background] Wexler D, Searles G, Landells I, Shear NH, Bissonnette R, Papp K, Poulin Y, Langley R, Gulliver WP. Update on alefacept safety. J Cutan Med Surg. 2009 Dec;13 Suppl 3:S139-47. doi: 10.2310/7750.2009.00032. PMID 20053326
- See also: Link to FDA Website — http://www.accessdata.fda.gov/scripts/cder/drugsatfda